CLINICAL TRIAL: NCT04802564
Title: Multisensory Biofeedback With Musical Interface for Sensorimotor Control Capacity of Hands
Brief Title: Musical Biofeedback for Sensorimotor Control Capacity of Hands
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: A-ER-108-557
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2024-11

CONDITIONS: Hand Injuries
Keywords: musical biofeedback; auditory; vibrotactile stimulation
MeSH Terms: conditions — Hand Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multisensory-based music treatment (Experimental): Using a multisensory-based music treatment synchronizing with vibrotactile stimulation on the finger pulps during the protection phase (week 0-4) for hand injury patients.
  Interventions: Other: regular hand therapy
- Traditional sensory reeducation intervention (Active Comparator): Using constant and moving tactile stimulation on the finger pulps during the protection phase (week 0-4) for hand injury patients.
  Interventions: Other: regular hand therapy

INTERVENTIONS:
Other: regular hand therapy — edema control, scar management, stretching regimen, tendon gliding exercise, blocking exercise, muscle strengthening protocols

SUMMARY:
In the proposed study, the investigators assumed that music support treatment, a multisensory-based framework for ameliorating brain plasticity, combined with low-amplitude vibration stimulation can prime motor system and change in motor performance for the patient with a peripheral injury or the loss of a limb. The specific aim of this study is to develop a Multisensory Biofeedback with Musical Interface system, with the aim of improving the sensorimotor impairment of patients' hands.The expected outcomes of this research are to clarify the effects of application Multisensory Biofeedback with Musical Interface on motor and hand function for patients with hand injuries.

ELIGIBILITY:
Inclusion Criteria:

* tendon and bone injury in hand, wrist, and forearm; peripheral nerve injury in upper extremity; replantation; a combination of nerve and tendon or vascular injury; the protective sensation of the hand is absent or impaired

Exclusion Criteria:

* patients with deficits in cognition, perception or language comprehension, as well as severe pain and swelling in the upper limbs

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2025-06-11 (Actual); Study Completion 2025-06-11 (Actual)

PRIMARY OUTCOMES:
Change in the result of pinch-holding-up-activity test | 8 weeks, 12 weeks and 24 weeks

SECONDARY OUTCOMES:
Chang in the result of two-point discrimination (S2PD) test | 4 weeks, 8 weeks, 12 weeks and 24 weeks
Chang in the result of Semmes-Weinstein monofilament (SWM) test | 4 weeks, 8 weeks, 12 weeks and 24 weeks
Chang in the result of active range of motion test | 4 weeks, 8 weeks, 12 weeks and 24 weeks
Change in the result of Purdue pegboard test | 8 weeks, 12 weeks and 24 weeks
Change in the result of Minnesota manual dexterity test | 8 weeks, 12 weeks and 24 weeks
Change in the result of Manual ability measurement | 4 weeks, 8 weeks, 12 weeks and 24 weeks
Change in the result of Near-Infrared Spectroscopy | 4 weeks and 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- National Cheng-Kung University Hospital, Tainan, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu HY, Lin CW, Lin YC, Wu PT, Kato H, Su FC, Kuo LC. Effects of vibrotactile-enhanced music-based intervention on sensorimotor control capacity in the hand of an aging brain: a pilot feasibility randomized crossover trial. BMC Geriatr. 2021 Nov 23;21(1):660. doi: 10.1186/s12877-021-02604-0. PMID 34814839